CLINICAL TRIAL: NCT05903196
Title: Study of the Use of Radiofrequency Ablation in LatinX Patients With Symptomatic Benign Thyroid Nodules
Brief Title: Radiofrequency Ablation Study in LatinX Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Daniel Kuriloff, Director, Center for Thyroid & Parathyroid Surgery, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0711
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mygen V-1000 RF system (Experimental): The Mygen V-1000, a microprocessor-based generator of RF Medical Co., Ltd., provides up to 140 watts of radio-frequency (RF) energy to be used for coagulation & ablation of vessel, tissue & bone
  Interventions: Device: Mygen V-1000 RF system

INTERVENTIONS:
Device: Mygen V-1000 RF system — The Mygen V-1000, a microprocessor-based generator of RF Medical Co., Ltd., provides up to 140 watts of radio-frequency (RF) energy to be used for coagulation & ablation of vessel, tissue & bone

SUMMARY:
Benign thyroid nodules can still create cosmetic, compressive, or hormonal issues for patients. In the past, surgery was typically used to treat thyroid nodules causing the above issues through partial or complete thyroidectomy. More recently, minimally-invasive techniques have been developed to treat these issues. This study is investigating the use of one of these techniques, radiofrequency ablation, in Latinx patients with benign symptomatic thyroid nodules. This procedure is of interest because it avoids the risks of surgery and can be done outside an operating room. The study hypothesis is that the use of RFA is an effective and safe therapeutic option for LatinX patients with a symptomatic benign nodule wishing to avoid surgery.

DETAILED DESCRIPTION:
Thyroid nodules can create issues for individuals such as affecting the level of their thyroid hormones, causing an unwanted physical appearance, or pressing on other important structures in the neck (for example, trachea and esophagus). In the past, surgery was typically used to treat thyroid nodules causing the above issues, either taking out some or all of the thyroid. More recently, new techniques that do not require surgery have been developed to treat these issues. This study is investigating the use of one of these newer techniques, called radiofrequency ablation in Latinx patients with non-cancerous symptomatic thyroid nodules. This procedure is of interest because it avoids the risks of surgery (like bleeding, infection, scars) and can be done in a clinic setting. The theory is that this procedure will be a safe and effective alternative to surgery for non-cancerous thyroid nodules that are causing symptoms in Latinx patients, which is a population in which this treatment has not yet been studied. Patients who decide to enroll in the study will be required to fill out questionnaires, have blood tests, have ultrasounds of the thyroid, and undergo the radiofrequency ablation minimally-invasive treatment instead of surgery. Patients will be evaluated at 1 month, 3 months, 6 months, 12 months, and 18 months after the procedure to assess for effectiveness of the procedure and any side effects.

Most evidence supporting RFA of thyroid nodules comes from international cohorts. In a recent meta-analysis, RFA accomplished volume reduction ranging from 68 to 87% in over 1100 treated nodules. This reduction was sustained for up to 5 years. In terms of its safety, a recent systematic review of 2700 nodules showed only 41 major complications and 48 minor complications from RFA. Of note, most complications were transient, only 4 patients developed permanent voice changes, while 1 required rescue lobectomy after a nodule ruptured. Published data in the United States also showed RFA to be an effective and safe strategy. However, of the 47 studied patients, none were LatinX. Furthermore, lack of coverage by insurance companies means this procedure is typically only available as an out-of-pocket expense and is therefore out of reach for underserved patients. Data to establish the safety/feasibility of this novel intervention is needed for the LatinX population.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Subjects over 18 years of age
* Subject who self-identifies as LatinX
* Subjects who have a benign, symptomatic thyroid nodule
* Subjects whose nodule has well-defined margin on ultrasound and is surrounded by at least 2mm of normal thyroid parenchyma in all directions

Exclusion Criteria:

* Patients who are pregnant, trying to become pregnant, or breastfeeding
* Patient who have a cardiac pacemaker,defibrillator , or other electromedical equipment
* Patients who have a nodule that is malignant or not predominantly solid (must be >50% solid by ultrasound)
* Patients who cannot give consent
* Patients on anticoagulation or dual antiplatelet therapy
* Patients with acute illness
* People with BP > 140/90 prior to the scheduled procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related changes in thyroid nodule volumes | 2 years
  To study the change in nodule volume

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kuriloff, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Physician Partners, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided